CLINICAL TRIAL: NCT04702789
Title: Phase IV Clinical Study to Compare the Efficacy of the Krytantek Ofteno PF® Plus Gaap Ofteno PF® Combination to the Krytantek Ofteno PF® Plus Gaap Ofteno PF® Combination, in Primary Open Angle Glaucoma or Ocular Hypertension Patients.
Brief Title: Comparative Study of the Efficacy of Either Krytantek Ofteno PF® or Eliptic Ofteno PF® Plus Gaap Ofteno PF® for POAG or Ocular Hypertension.
Acronym: PRO-122
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: For interests of sponsor.
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH122-0420/IV
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost; dorzolamide-timolol combination

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, multicenter with parallel groups.
Who Masked: Participant, Investigator
Masking Description: After signing the informed consent form (ICF), every subject will receive a coded patient number. Randomization will take place through and integrated web response system (IWRS). In the first step, during the eligibility visit, all patients will be assigned the same treatment (Gaap Ofteno PF®). After one month, patients that once again comply with the inclusion criteria will be assigned randomly (1:1) to one of the two investigation products, either Krytantek Ofteno PF® or Eliptic Ofteno PF®.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1; Dorzolamide-timolol-brimonidine and latanoprost; Krytantek Ofteno PF® and Gaap Ofteno PF® (Experimental): Application of Gaap Ofteno® (latanoprost 0.005%; preservative free) ophthalmic solution every 24 hours at 21:30 hours (± 15 min) for the duration of the study (total exposure: 90 days). One month after initiating Gaap Ofteno® instillation, application of Krytantek Ofteno® (dorzolamide 2%, timolol 0.5% and brimonidine 0.2%; preservative free) ophthalmic solution will be added every 12 hours at 9:00 and 21:00 hours (± 10 min) (total exposure: 60 days).
  Interventions: Drug: Dorzolamide-timolol-brimonidine and latanoprost
- Arm 2; Dorzolamide-timolol and latanoprost; Eliptic Ofteno PF® and Gaap Ofteno PF® (Experimental): Application of Gaap Ofteno® (latanoprost 0.005%; preservative free) ophthalmic solution every 24 hours at 21:30 hours (± 15 min) for the duration of the study (total exposure: 90 days). One month after initiating Gaap Ofteno® instillation, application of Eliptic Ofteno® (dorzolamide 2% and timolol 0.5%; preservative free) ophthalmic solution will be added every 12 hours at 9:00 and 21:00 hours (± 10 min) (total exposure: 60 days).
  Interventions: Drug: Dorzolamide-timolol and latanoprost

INTERVENTIONS:
Drug: Dorzolamide-timolol-brimonidine and latanoprost — Application of Gaap Ofteno PF® every 24 hrs for 30 days plus concomitant application of Krytantek Ofteno PF® every 12 hours for 60 days. Total intervention time: 90 days.
  Other Names: PRO-122; Krytantek Ofteno PF®; Gaap Ofteno PF®
  Arms: Arm 1; Dorzolamide-timolol-brimonidine and latanoprost; Krytantek Ofteno PF® and Gaap Ofteno PF®
Drug: Dorzolamide-timolol and latanoprost — Application of Gaap Ofteno PF® every 24 hrs for 30 days plus concomitant application of Eliptic Ofteno PF® every 12 hours for 60 days. Total intervention time: 90 days.
  Other Names: Eliptic Ofteno PF®; Gaap Ofteno PF®
  Arms: Arm 2; Dorzolamide-timolol and latanoprost; Eliptic Ofteno PF® and Gaap Ofteno PF®

SUMMARY:
Phase IV randomized, double blind, multicenter, parallel group clinical study to evaluate the efficacy of the combined use of Krytantek Ofteno PF® and Gaap Ofteno PF®, both applied every 12 hours, versus the use of Eliptic Ofteno PF® Plus Gaap Ofteno PF®, both applied every 12 hours, in patients with open angle glaucoma or ocular hypertension during 90 days

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed primary open angle glaucoma or ocular hypertension, not using a prostaglandin analogue or a β-blocker in the eye to be included in this study.
* No treatment with any prostaglandin analogues or a β-blockers within the 30 days previous to eligibility visit, in the eye to be included in this study.
* IOP measured with Goldmann tonometer ≥ 19 and ≤ 26 mmHg, in the eye to be included in this study.
* Being capable of voluntarily grant a signed informed consent.
* Being willing and able to meet the requirements of the study such as attending programmed visits, treatment plan and other study procedures.
* Age ≥18 years old.

Exclusion Criteria:

* Pregnancy, breastfeeding or planning to become pregnant during the time of the study
* In the case of women of childbearing age, not counting with a hormonal contraceptive method, intrauterine device or bilateral tubal obstruction.
* Anterior chamber angle < 2 in Shaffer's scale, or presence of peripheral anterior synechia, in the eye to be included in the study.
* Being currently under treatment with any systemic ocular hypotensive drug (mannitol, glycerin, isosorbide, etc).
* BCVA worse than 20/200, in the eye to be included in the study.
* Serious loss of central visual field (sensibility ≤ 10 dB in ≥ 2 of the central sites), in the eye to be included in the study.
* Having a previous history of any ophthalmological surgical or laser procedure, within the last 6 months, in the eye to be included in thee study.
* Previous history of ocular trauma within the last 6 months, in the eye to be included in thee study.
* Previous history of chronic uveitis, in the eye to be included in the study.
* Previous history of intraocular, periocular, retrobulbar, subconjunctival or sub-tenon injection within the last 6 months, in the eye to be included in the study.
* Patients with or that have had silicone present in either the anterior or posterior segments of the eye to be included in the study.
* Aphakia in the eye to be included in the study.
* Presence of any corneal alteration that may decrease the reliability of Goldmann tonometry in the eye to be included in the study.
* Known hypersensitivity to any of the active principles to be used in the study (prostaglandin analogues, β-blockers, α2-agonists, carbonic anhydrase inhibitors).
* History of any disease that contraindicates the use of the active principles to be used in the study (asthma, chronic obstructive pulmonary disease (COPD), 2nd or 3rd degree auriculoventricular blockade without pacemaker, sinus bradycardia, manifest cardiac insufficiency, chronic kidney disease with a creatinine clearance < 30 ml/min).
* Requirement of use of monoamineoxidase inhibitors and patients using antidepressants that affect noradrenergic transmission (tricyclic antidepressants and mianserin).
* Patients who use, or have used within the las month, steroids applied topically in the eye to be included in the study or through oral, intravenous, intramuscular, dermic, or intralesional administration.
* Having participated in clinical trials within 30 days prior to signing this study's informed consent form.
* Having participated previously in this study.
* Previous history of drug addiction within the last 2 years prior to signing this study's informed consent form.
* Having any kind of programmed surgery during the period of this study.
* Being or having any immediate family members (spouse, parent/legal tutor, sibling or child) who work either in the investigation center or for the sponsor of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Change in intraocular Pressure (IOP) | Days: -30 (± 2) (eligibility visit), 0 (basal visit), 14 (± 2) (first follow-up visit), 30 (± 2) (second follow-up visit) and 60 (± 2) (final visit)
  Measured through Goldman tonometer in milligrams of mercury (mmHg). After instillation of topical anesthetic (tetracaine 0.5%) and fluorescein stain, IOP is evaluated at 9:00 and at 11:00 hrs. (± 30 minutes). Both measurements and their average will be registered. Normal values are considered between 10 and 21 mmHg.

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) | Days: -30 (± 2) (eligibility visit), 0 (basal visit), 14 (± 2) (first follow-up visit), 30 (± 2) (second follow-up visit) and 60 (± 2) (final visit)
  With the patient's best possible refractive correction, visual acuity will be evaluated through the Snellen chart. Its notation (fraction or decimal) is described as the distance from the chart at which the test is performed, divided by the distance at which a letter equals vertically 5 minutes of arc.
Changes in optic nerve cup/disc ratio | Days: -30 (± 2) (eligibility visit), 0 (basal visit) and 60 (± 2) (final visit)
  Both clinical and imaging evaluation will be performed. For clinical evaluation, after the application of a topical ophthalmic mydriatic (tropicamide 0.8% / phenylephrine 5%), indirect ophthalmoscopy will be performed through the aid of a fundus lens in a slit lamp. For imaging, optic coherence tomography (OCT) will be used.
Change in nerve fibers and ganglion cell thickness | Days: 0 (basal visit) and 60 (± 2) (final visit)
  Spectral domain OCT is a non invasive tool that will be used to evaluate quantitatively the thickness of retinal nerve fibers and ganglion cell layers.
Change in optic nerve image | Days: -30 (± 2) (eligibility visit), 0 (basal visit) and 60 (± 2) (final visit)
  Through a fundus camera a photograph will be taken to obtain a faithful record of any possible changes to the optic nerve head characteristics.
Change in central corneal thickness | Days: 0 (basal visit) and 60 (± 2) (final visit)
  Measured through ultrasonic pachymetry, three assessments will be performed, these and its average will be recorded.
Change in visual fields | Days: 0 (basal visit) and 60 (± 2) (final visit)
  Visual fields will be evaluated with a SITA standard automated white-on-white perimetry performed with a Humphrey perimeter. To be considered reliable, fixation losses, false positives and false negatives must be under 20%. Mean deviation (MD) and pattern standard deviation (PSD) will be recorded.
Change in ocular surface integrity (conjunctival hyperemia, chemosis, and corneal fluorescein staining) | Days: -30 (± 2) (eligibility visit), 0 (basal visit), 14 (± 2) (first follow-up visit), 30 (± 2) (second follow-up visit) and 60 (± 2) (final visit)
  By means of a slit lamp, conjunctival hyperemia, chemosis, and corneal fluorescein staining will be evaluated. Conjunctival hyperemia will be graded according to Efron's scale (5 grades: Normal (0), Very Mild (I), Mild (II), Moderate (3), and Severe (4)). Chemosis will be evaluated as present (if conjunctiva separates from the sclera in ≥ 1/3 of the palpebral opening area or if it exceeds the eyelid's gray line) or absent. Fluorescein staining evaluation will take place after applying the fluorescein stain on the ocular surface and evaluating the resulting staining pattern. This will be measured through the Oxford scale which includes 6 grades: Absent (0), Minimal (I), Mild (II), Moderate (III), Marked (IV), Severe (V).
Incidence of adverse events | Day: 75 (± 3) (safety call)
  Presence/absence adverse events, defined as the appearance of any unfavorable reaction in a patient participating in a clinical investigation in which any pharmaceutical product is being administered, regardless of the causal attribution.
Changes in Ocular Comfort Index | Days: -30 (± 2) (eligibility visit), 0 (basal visit), 14 (± 2) (first follow-up visit), 30 (± 2) (second follow-up visit) and 60 (± 2) (final visit)
  Ocular Comfort Index (OCI) Questionnaire will be used for evaluation of tolerability through incidence and severity of dry eye symptoms in a scale from 0 to 100. Greater scores mean a worse outcome.

OTHER OUTCOMES:
Proportion of patients who reached a specific IOP decrease in mmHg | Days: 60 (± 2) (final visit)
  Patients who reached IOP within the following ranges: ≤12, ≤13, ≤14, ≤15, or ≤18.
Proportion of patients who reached a specific IOP decrease in percentage | Days: 60 (± 2) (final visit)
  Patients who demonstrated decrease in IOP within the following percentage ranges: ≥ 20%, ≥ 25%, ≥ 30%, y ≥ 35%

CONTACTS AND LOCATIONS:
Locations (1):
- Servicios Médicos y de Investigación Clínica InspirePharma S. de R.L.de C.V., Monterrey, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olvera-Montano O, Mejia-Morales C, Jauregui-Franco RO, Gomez-Mendez SC, Munoz-Villegas P. Maximum Tolerated Medical Therapy for Glaucoma: Fixed-Dose Combinations of Timolol, Dorzolamide, Brimonidine with Latanoprost Versus Timolol, Dorzolamide with Latanoprost. Clin Ophthalmol. 2025 Aug 22;19:2913-2925. doi: 10.2147/OPTH.S540312. eCollection 2025. PMID 40873654